CLINICAL TRIAL: NCT07193745
Title: Respiratory Function, Functional Capacity, Physical Activity, and Fatigue in Patients With Systemic Lupus Erythematosus: A Cross-Sectional Study
Brief Title: Respiratory Function, Physical Activity and Fatigue in SLE
Status: Recruiting | Type: Observational
Sponsor: Melis Usul (Other)
Responsible Party: Sponsor-Investigator, Melis Usul, Specialist Physiotherapist, Istanbul Kent University
Organization: Istanbul Kent University (Other)
Other Study IDs: 2025/05-1560
Record Dates: First submitted 2025-09-15; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: respiratory function; functional capacity; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with systemic lupus erythematosus: Individuals diagnosed with systemic lupus erythematosus according to the American College of Rheumatology classification criteria. Participants will be adults aged 18-65 years.
- Healthy individuals: Age- and sex-matched healthy participants without any medical conditions (including neurological, genetic, or psychiatric disorders) that would prevent them from completing the tests.

SUMMARY:
Increasing awareness of possible pulmonary involvement in patients with systemic lupus erythematosus (SLE) will enable earlier diagnosis of the disease and minimize damage accumulation. According to our research, no study has been found that examines respiratory functions in detail in SLE patients and investigates their relationship with functional capacity, physical activity, and fatigue levels. Our primary aim is to compare respiratory functions, functional capacity, physical activity, and fatigue levels between patients with SLE and healthy controls. Our secondary aim is to investigate the relationship between respiratory functions with functional capacity, physical activity levels, and fatigue in SLE patients.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic, inflammatory, autoimmune disease characterized by multisystem involvement. SLE can affect any organ or tissue, including the skin, joints, kidneys, central and peripheral nervous systems, lungs, and heart. Approximately 50% of patients with SLE may experience pulmonary involvement during the course of their disease. The most commonly reported manifestations in patients with SLE are pleurisy, diffuse alveolar hemorrhage, shrinking lung syndrome, interstitial lung disease, and pulmonary arterial hypertension.

Although estimates exist, the exact prevalence of pulmonary disease is unknown, and study findings have varied. In this context, our aim is to compare respiratory function, functional capacity, physical activity, and fatigue levels in patients with SLE with those in healthy controls. Our secondary aim is to investigate the relationship between respiratory function and functional capacity, physical activity level, and fatigue in patients with SLE.

Pulmonary function of the patients will be evaluated using pulmonary function tests. The level of physical activity of the participants will be assessed using the Global Physical Activity Questionnaire. Functional capacity will be evaluated with the 6-Minute Walk Test. Fatigue will be assessed using the Fatigue Severity Scale. Statistical analyses of the data obtained from the study will be performed using the Statistical Package for Social Sciences (SPSS) software.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been followed with a diagnosis of systemic lupus erythematosus for at least 1 year
* Able to ambulate independently
* No cognitive or mental impairment
* Willing to participate in the study

Exclusion Criteria:

* Presence of major musculoskeletal disease affecting the lower extremities
* Presence of severe disease affecting the cardiovascular system
* Being pregnant
* Smoking
* Having a diagnosis of restrictive/interstitial lung disease due to the underlying condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-65 years with a diagnosis of SLE
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | Time Frame: Baseline (day of enrollment) assessment
  The pulmonary function test will be performed using the COSMED Pony FX device in accordance with the American Thoracic Society and European Respiratory Society guidelines.
Forced Expiratory Volume (FEV1) | Baseline (day of enrollment) assessment
  The pulmonary function test will be performed using the COSMED Pony FX device in accordance with the American Thoracic Society and European Respiratory Society guidelines.
Tiffeneau Index (FEV1/FVC) | Baseline (day of enrollment) assessment
  The pulmonary function test will be performed using the COSMED Pony FX device in accordance with the American Thoracic Society and European Respiratory Society guidelines.
Peak Expiratory Flow (PEF) | Baseline (day of enrollment) assessment
  The pulmonary function test will be performed using the COSMED Pony FX device in accordance with the American Thoracic Society and European Respiratory Society guidelines.
Functional Capacity | Time Frame: Baseline (day of enrollment) assessment
  Functional capacity is assessed using the 6-Minute Walk Test according to the criteria of the American Thoracic Society. Participants are instructed to walk as fast as possible, but without running, at their own pace along a 30-meter flat corridor for 6 minutes. The distance covered is recorded in meters.
Physical Activity Level | Baseline (day of enrollment) assessment
  The participants' physical activity status is assessed using the Global Physical Activity Questionnaire. The questionnaire consists of 16 questions. In the work and leisure activity sections, vigorous and moderate physical activities are assessed, while in the transportation section, moderate physical activities are assessed. In addition, there is an extra question for sedentary time. In each section, one yes/no question is followed by open-ended questions on the number of days per week and the duration per day. As a result of the questionnaire, the total weekly MET-minutes of physical activity are calculated. Moderate-intensity physical activities correspond to 4 MET/min, and vigorous-intensity physical activities correspond to 8 MET/min. Weekly total MET-minutes are calculated by multiplying with these coefficients.

SECONDARY OUTCOMES:
Fatigue Level | Baseline (day of enrollment) assessment
  Fatigue is assessed using the Fatigue Severity Scale. The scale consists of 9 items. Participants are asked to select a number from 1 to 7 for each statement, indicating the extent to which they agree with it (1: strongly disagree; 7: strongly agree). The scores obtained for all items are summed and then divided by nine to calculate the final score. A score of four or higher generally indicates severe fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Ela Tarakçı, Professor, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No